CLINICAL TRIAL: NCT04530695
Title: Early Diagnosis and Treatment of Periodontal Disease in Patients With AML to Reduce Bloodstream Infections During Chemotherapy
Brief Title: Diagnosis and Treatment of Periodontal Disease in Patients With AML
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution and research was cancelled due to his departure
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020LS118
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: AML; Acute Myelogenous Leukemia
Keywords: AML; Periodontitis; Blood stream infections
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Deep Cleaning (Experimental): participants with periodontitis will undergo treatment by scaling and root planing (SRP)
  Interventions: Other: Scaling and Root Planing
- Arm B: No cleaning (No Intervention): participants with periodontitis will undergo no periodontal treatment

INTERVENTIONS:
Other: Scaling and Root Planing — Periodontal treatment by scaling and root planing (SRP), deep cleaning
  Other Names: SRP
  Arms: Arm A: Deep Cleaning

SUMMARY:
This is a phase 2 randomized controlled trial of pre-chemotherapy periodontal deep cleaning in Acute Myelogenous Leukemia (AML) patients with asymptomatic periodontitis.

Once eligibility is confirmed, participants with periodontitis will be randomized in a 1:1 ratio to undergo treatment by scaling and root planing (SRP, "deep cleaning") (arm A) or receive no periodontal treatment (arm B). We will compare the incidence of Blood Stream Infection (BSI) during chemotherapy between the two arms.

Study participation will continue until day 28 of chemotherapy or discharge from hospital, whichever occurs first.

DETAILED DESCRIPTION:
Bloodstream infection (BSI) is common in patients with acute myeloid leukemia (AML) and causes significant morbidity and mortality. Chemotherapy disrupts oral and intestinal mucosal barriers, facilitating bacterial translocation to the bloodstream.

Baseline periodontitis is associated with higher risk of BSI during chemotherapy. In AML patients, since baseline screening and treatment of asymptomatic periodontitis is currently not a standard practice, the researchers are hoping to (i) personalize supportive care according to patient-specific risk factors; (ii) promote an interdisciplinary approach to supportive care by bringing periodontists into the treatment team; (iii) improve quality of life by reducing hospitalization length; (iv) decrease the incidence of re-hospitalization during future phases of treatment; (v) decrease early treatment related mortality (TRM); and (vi) decrease healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Newly diagnosed or relapsed AML
* Planned intensive chemotherapy (Any regimen expected to require 3-4 weeks of inpatient stay)
* Antibacterial prophylaxis using levofloxacin 500 mg daily
* Sufficient time to perform periodontal examination and treatment by day 1 of chemotherapy

Exclusion Criteria:

* Prior treatment for AML, except hydroxyurea or leukapheresis
* ANC <0.5 x 10^9/L at the time of enrollment
* Post-transfusion platelet count <50x10^9/L at the time of enrollment
* Unstable for transfer to the School of Dentistry
* Fever at the time of enrollment
* Documented infection at the time of enrollment
* SRP in the last 3 months
* Symptomatic periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of neutropenic fever (NF) by day 28 of chemotherapy or discharge | Day 28 or discharge date (whichever occurs first)

SECONDARY OUTCOMES:
Incidence of BSI by day 28 of chemotherapy or discharge | Day 28 or discharge date (whichever occurs first)
  Incidence of bloodstream infections by day 28 of chemotherapy or discharge (whichever occurs first).
Incidence of blood culture-negative NF by day 28 of chemotherapy or discharge, whichever occurs first | Day 28 or discharge date (whichever occurs first)
Incidence of oral mucositis by day 28 of chemotherapy or discharge, whichever occurs first | Day 28 or discharge date (whichever occurs first)
Incidence of death by day 28 | Day 28 or discharge date (whichever occurs first)
Number of days hospitalized | Upto 8 weeks
  Hospitalization length
Incidence of Neutropenic Fever within 2 days after periodontal examination/treatment (safety endpoint) | within 2 days after periodontal examination/treatment

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — University of Minnesota, Division of Hematology, Oncology and Transplantation